CLINICAL TRIAL: NCT07113860
Title: Reframing Expectations About Aging - Physical Activity and Inclusive Reappraisal (RE-PAIR): Protocol of an Intervention Aiming to Promote Positive Views on Aging and Behavior Change in Older Couples
Brief Title: Reframing Expectations About Aging - Physical Activity and Inclusive Reappraisal
Acronym: RE-PAIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Catholic University of the Sacred Heart (Other); Ecole Normale Supérieure de Rennes (Unknown); University of Padova (Other); University of Kaiserslautern-Landau (Other); Flinders University (Other); University of Greifswald (Other); Federico II University (Other); North Carolina State University (Other); Humboldt-Universität zu Berlin (Other)
Responsible Party: Principal Investigator, Serena Sabatini, PhD in Psychology, University of Barcelona
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: LCF/BQ/PI24/12040008
Record Dates: First submitted 2025-07-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Self-perceptions of Aging; Physical Activity
Keywords: Physical activity; Walking; Self-Perceptions of Aging; Ageism; Subjective aging; couples; spouses
MeSH Terms: conditions — Motor Activity; Ageism

STUDY DESIGN:
Intervention Model Description: In the first group/arm, both partners/spouses will undertake the intervention together. In the second group/arm, only one of the two partners will undertake the intervention during data collection. In the third (control) group/arm none of the partners will undertake the intervention during data collection.
Who Masked: Outcomes Assessor
Masking Description: The person who will interact with participants to send out questionnaires, plan assessment dates, etc will be blinded. The person who assesses participants will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention delivered to both partners/spouses (Experimental): Both partners/spouses will undertake together a multi-component intervention comprising a psychoeducational component (aiming to promote positive views on aging via three in-person sessions) and a behavioral component (asking participants to start walking up to five times per week for 12 weeks).
  Interventions: Behavioral: Views on Aging Intervention; Behavioral: Projecte Moviment
- One partner/spouse undertakes the intervention (Active Comparator): Only one of the two partners/spouses will undertake the multi-component intervention during data collection. The remaining partner will be offered the opportunity to undertake the intervention at the end of data collection. The intervention is the same delivered to arm one and it comprises a psychoeducational component (aiming to promote positive views on aging via three in-person sessions) and a behavioral component (aiming to promote walking up to five times per week for 12 weeks).
  Interventions: Behavioral: Views on Aging Intervention; Behavioral: Projecte Moviment
- Partners/spouses do not undertake the intervention (No Intervention): This is the control group/arm. None of the spouses/partners undertakes the intervention during data collection. They will be offered the opportunity to undertake the intervention at the end of data collection.

INTERVENTIONS:
Behavioral: Views on Aging Intervention — This intervention was developed by Wolff, Warner (47) in 2013-2014; refined by Beyer, Wolff (59) in 2017-2018; and further refined for this project. It will be delivered through three in-person one-hour sessions by two psychologists. it will include homework between sessions two and three. The first session will consist of a quiz on aging with questions about healthy aging and aging in general to detect own negative personal views on aging and misconceptions regarding aging. The second session will provide information on the benefits of more positive views on aging on health, functional and cognitive abilities, and longevity. During the third session participants are thought a technique to modify negative automatic thoughts about aging and asked/invited to put in practice this technique. Finally, the intervention ends with a focus on positive views on aging and their importance for one's health and wellbeing.
  Arms: Intervention delivered to both partners/spouses; One partner/spouse undertakes the intervention
Behavioral: Projecte Moviment — The intervention lasts 12 weeks and is based on international guidelines of physical exercise. Participants will be instructed to walk briskly in one continuous bout (45 minutes for 5 days, 225 minutes per week). Intensity, duration, and times per week will be initiated in a stepwise manner to reduce the possibility of injury. During the first week participants will be asked to walk 30 minutes at 9-10 on the Borg Rating of Perceived Exertion Scale (i.e., light intensity). During the second week, participants will be asked to walk 45 minutes with the same intensity. During the remaining weeks, participants will be asked to maintain the duration of 45 minutes and increase the intensity of the activity to a moderate-high effort that corresponds with 12-14 in the Borg Rating of Perceived Exertion Scale.
  Arms: Intervention delivered to both partners/spouses; One partner/spouse undertakes the intervention

SUMMARY:
The goal of this clinical trial is to promote positive views on aging and walking in Spanish partners aged 65 years and over. The trial will comprise three arms. In the first arm, both partners will undertake the intervention together. In the second arm, only one of the two partners will undertake the intervention. In the third arm (control) none of the partners will undertake the intervention. Collection of quantitative data will make it possible to test the following hypotheses:

1. Differently from arm three, those participants from arms one and two who undertake the intervention will experience changes in primary and secondary intervention outcomes between pre- and post-intervention and these changes will be maintained at follow-ups.
2. Compared to delivering the intervention to only one partner, delivering it to both partners will lead to a greater and more lasting change in primary and secondary intervention outcomes.
3. In the group where only one partner will undertake the intervention, their change in intervention outcomes is observed at least to a small extent in the other partner.

Qualitative data collected at the end of the intervention through interviews of ten couples from each of arms one and two will make it possible to test three additional research questions:

1. How do participants in Group one engage with the intervention tasks, and to what extent do they undertake these tasks jointly as a couple?
2. In what ways do participants in Group two involve their non-participating partner in the intervention activities?
3. What changes do participants in Groups one and two report in their views of themselves and their aging, as well as in their perceptions of and interactions with their partner?

Participants will undertake a multicomponent intervention comprising:

* Three in-person psychoeducational sessions aiming to promote positive views on aging, including positive self-perceptions of aging, and accurate facts about aging
* Independent walking for 12 weeks Primary intervention outcomes are changes in participants' self-perceptions of aging and physical activity engagement. Secondary intervention outcomes are changes in ageism, subjective views of couple's joint aging, perceived age-related changes in one's partner, mood, physical fitness, and cognitive functioning.

DETAILED DESCRIPTION:
The current study will adopt a randomized pre- and post- intervention/trial design. A multicomponent (psychoeducational and behavioral) intervention called RE-PAIR (Reframing Expectations about aging - Physical Activity and Inclusive Reappraisal) and aiming to promote positive self-perceptions of aging and walking in older couples (i.e., spouses, cohabiting partners, or long-standing non-cohabiting partners) will be delivered to three intervention arms. In the first arm, both partners will undertake the intervention together. In the second arm, only one of the two partners will undertake the intervention. In the third (control) arm none of the partners will undertake the intervention.

Quantitative data collected through this trial design will make it possible to test four main hypotheses. First, based on previous research that tested the efficacy of the same psychoeducational intervention that will be used in this trial, it is hypothesized that, differently from the control group, those participants who undertake the intervention will experience changes in primary and secondary intervention outcomes between pre- and post-intervention and these changes will be maintained at follow-ups. Primary intervention outcomes are changes in self-perceptions of aging and physical activity engagement. Secondary intervention outcomes are changes in ageism, subjective views of couple's joint aging, perceived age-related changes in one's partner, mood, physical fitness, and cognitive functioning. Second, based on previous evidence on physical activity, it is hypothesized that compared to when delivering the intervention to only one partner, delivering it to both partners will lead to a greater and more lasting change in primary and secondary intervention outcomes. Third, it is hypothesized that in the group/arm where only one partner will undertake the intervention, their change in intervention outcomes is observed at least to a small extent in the other partner due to partners tending to influence each other's beliefs and behaviors. Finally, qualitative data collected at the end of the intervention through interviews of ten couples from each of groups 1 and 2 will make it possible to test three additional research questions. First, how do participants in arm 1 engage with the intervention tasks, and to what extent do they undertake these tasks jointly as a couple? Second, in what ways do participants in arm 2 involve their non-participating partner in the intervention activities? Third, what changes do participants in arms 1 and 2 report in their views of themselves and their aging, as well as in their perceptions of and interactions with their partner?

After having obtained participants' written informed consent in person, baseline, immediately post-intervention, and six-month follow-up assessments will be conducted as one-on-one sessions in the facilities of the Department of Clinical Psychology and Psychobiology of the University of Barcelona or in collaborating centers. During these assessments, participants will also independently complete some online questionnaires. The three-month follow-up assessment will instead be conducted online only. The sessions of the psychoeducational intervention will be conducted as group sessions in a small seminar room of the Department of Clinical Psychology and Psychobiology at the University of Barcelona or in collaborating centers. The behavioral component of the intervention will be undertaken independently by participants after having received instructions by the researchers.

This study aims to recruit 342 participants (i.e., 171 couples), randomly allocating 114 (i.e., 57 couples) to each of the three intervention arms. It is estimated that 342 participants are needed to provide 90% power at the two-sided 5% level of significance to detect a mean change of three units (i.e., moderate effects) on personal views on aging between any of the three study groups. As some participants may withdraw from the trial, the sample size calculation accounts for 30% drop out of participants.

It is expected that recruitment will last at least 12 months (between July 2025 and July 2026). Participants will be recruited via flyers, newsletters, and presentations at local organizations such as Amics de la Gent Gran; Fundació Catalunya La Pedrera; Universitat de l'experiència within the University of Barcelona; Federacio d'associacions de gent gran de Catalunya; IDIAP Jordi Gol Fundació Institut Universitari per a la Recerca a l'Atenció Primària de Salut Jordi Gol i Gurina. Primary care centers will also be contacted to recruit participants. Presentations will be delivered by the principal investigator (Dr Serena Sabatini) and a PhD candidate in Psychology. Participants will also be recruited through social media such as X, Facebook, Instagram, and LinkedIn. Snowballing technique will also be used. Should recruitment be slow, sources of recruitment will be diversified through contact of associations outside Barcelona.

Data collection is expected to start in September 2025 and to end at the end of April 2027. Those who fulfil inclusion criteria will be invited to take part in the study via email, phone text, and/or phone call. Baseline assessment will comprise an in-person assessment of 60 minutes at the University of Barcelona (or collaborating centers) and an online survey created using Microsoft forms. Starting from the in-person assessment, the researcher will first go through the information sheet with the participant and will ask the participant to report their informed written consent (about 10 minutes). Second, participants will undertake paper and pencil cognitive tasks (about 10 minutes). Third, participants will undertake a 15-minute physical fitness test. Fourth, using a computer facilitated by the researcher, participants will be asked to complete the first part of an online survey comprising questions on sociodemographic information, their physical health, their mood, their engagement in physical activities, social network, loneliness, intergenerational contact, and aspects of their relationship with their partner (taking approximately 25 minutes). Participants will then be asked to complete within 24 hours the second part of the online survey comprising questions about self-perceptions of aging; ageism; subjective views of couple's joint aging; personality traits; quality of marriage; and perceived age-related changes in one's partner (taking about one hour). Couples will then be randomly allocated by the principal investigator to one of the three intervention arms using a statistical software (i.e., STATA). Everyone from arm 1 and half of arm 2 (one partner per couple) will undertake the intervention at the University of Barcelona or at collaborating centers. Individuals of arm 1 will be assigned to the same intervention class of their partner. More specifically, arm 1 will be further divided into nine classes. Those from arm 2 who will undertake the intervention will be further divided into five classes. The partner from arm 2 who will receive the intervention will be randomly selected while taking into account for age and sex. As the control group will not receive an alternative intervention, participants will not be blinded with regard to group allocation. The control group will purposefully not receive an alternative intervention as this study aims to test the effects of the intervention compared to undertaking none. Moreover, the study team aims to undertake additional analyses in the control group/arm that will address research questions separate from this intervention study. During the 12-week intervention, participants who will receive the intervention will be asked to record in a-priori form every time they engage in physical activity. In doing so participants will also have to record how much and at which intensity - using the Borg Rating of Perceived Exertion Scale - they engaged in physical activity. During the last session of the in-person intervention participants will be asked to complete a paper and pencil questionnaire comprising a mix of multiple answers and open-ended questions (18 questions taking about 15 minutes). All participants (arms 1, 2, and 3) will be assessed again both in person and through self-administered online questionnaires at post-intervention and at six-months follow-ups. All participants will also be assessed through self-administered online questionnaires at three-month follow-up. In person they will complete the same cognitive tasks and physical fitness tests as at baseline assessment. Online they will complete a selection of baseline questionnaires assessing eventual changes in demographic information and physical health; general and personal views on aging; engagement in physical activities; ageism; subjective views of couple's joint aging; quality of marriage; and perceived age-related changes in their partner. In the two weeks following the last session of the intervention ten couples from arm 1 and ten couples from arm 2 will also undertake a 20-minute online interview using Phone/Teams/Zoom. Partners will be interviewed separately. Once data collection has ended, the remaining half of arm 2 and everyone from arm 3 will be offered the intervention as a big group.

The following measures will be used. Primary intervention outcomes

* Self-perceptions of aging: Awareness of Age-Related Change questionnaire, a one-item question assessing Felt Age, and a single-item assessing participants' Subjective Stage of Life.
* Self-reported physical activity will be assessed with the International Physical Activity Questionnaire short form and the Saltin-Grimby Physical Activity Level Scale.

Secondary intervention outcomes

* Experienced ageism will be assessed with the 15-item World Health Organization-Ageism Scale.
* Other directed-ageism over the past 12 months will also be assessed with nine additional questions developed by the Word Health Organization.
* Subjective views of couple's joint aging will be assessed with the 14-item Subjective Views of Couple's Joint Aging (SVoCJA).
* Mood will be assessed with the four-item version of the Patient Health Questionnaire (PHQ-4).
* Objective indicators of physical fitness will be body mass index, grip strength, and the Senior Fitness Test.
* Cognitive flexibility will be assessed with the paper and pencil version of the Trial Making Test.
* Working memory will be assessed with the paper and pencil version of the Digit Span Forward and Backward tasks taken from the Wechsler Adult Intelligence Scale, the PMR Phonological Verbal Fluency test, and the Animal Naming Fluency test.
* Sociodemographic questions will comprise age in years; sex; gender; sexual orientation; ethnic origin; highest level of education achieved and years of education; marital status; employment status; and total income. Participants will also fill the MacArthur's Scale of Subjective Social Status.
* Participants will be asked whether they have ever been diagnosed with a list of 21 chronic physical health conditions such as stroke and diabetes and with a list of 15 mental health conditions including depressive and anxiety disorder.
* The Ten-Item-Personality Inventory will be used to assess five personality traits: extraversion, agreeableness, openness, conscientiousness, and neuroticism.
* Quality of the relationship with one's partner will be assessed with the six-item Quality of Marriage Index.
* Dominance will be assessed using a single-item question: In your current romantic relationship, which one of you is more dominant/powerful? Participants will also be asked how many years they have been with their partner, whether they have children, and whether they have grandchildren.
* End-of-intervention questionnaire. At the end of the last intervention session all participants will complete, using pen and paper, a questionnaire comprising 18 between multiple answer and open-ended questions. These will assess perceived efficacy of the intervention, enjoyability of the intervention, and couple dynamics.
* Interviews. In the two weeks following the end of the in-person psychoeducational intervention, ten couples from intervention arm 1 and ten couples from intervention arm 2 will be randomly selected for online interviews via Phone/Teams/Zoom. Partners will be interviewed separately. Those participants who will have undertaken the intervention, will be asked to further elaborate on their answers on the end-of-intervention questionnaire. Those who will not have undertaken the intervention will be asked whether and how changes in their partner affected them.

Intervention Psychoeducational component targeting personal and general views on aging. The psychoeducational component of the intervention was developed by Wolff, Warner in 2013-2014 and further refined by Beyer, Wolff in 2017-2018 and proved effective at trial level in German older adults aged 66-88 years. In this project the intervention will be delivered through three in-person one-hour sessions delivered by two psychologists that will be different from the researchers/psychologists who will assess participants at baseline and follow-ups. The intervention will include homework between sessions two and three. To ensure comparability of content and procedure for all intervention groups, a modified version of Bayer and colleagues' 2019 intervention manual adapted for the Spanish population will be used. The first intervention session will consist of a quiz on aging with questions about healthy aging and aging in general to detect own negative personal views on aging as well as misconceptions regarding age and aging. Possible false beliefs will be corrected by providing information on empirical findings during the discussion of the answers. The second intervention session will occur three weeks later, and it will provide information on benefits of more positive personal views on aging regarding health, functional and cognitive abilities, as well as longevity. It will also include a group discussion on these benefits. Additionally, participants are given homework for the next intervention session. As part of the homework participants will be asked to observe themselves or others to detect negative age stereotypes or personal views on aging in everyday life and to write down the situations and the negative personal views on aging on a worksheet. At intervention session three, the homework will be presented and discussed in the group. Subsequently, a technique to change negative automatic thoughts about aging will be taught using a hypothetical situation. The technique consists of three steps: (1) sensitizing and increasing awareness of one's automatic and negative thoughts about aging, (2) questioning these thoughts and, (3) in the case of too negative thoughts, replacing them with more realistic, neutral, and/or more positive ones. To achieve steps two and three, participants will be asked to find some alternative, positive or neutral, and conceivable interpretations of the situation described. Finally, the intervention will end with a group discussion and by asking participants to write down some positive views on aging which are subsequently discussed in the group.

Behavioral component promoting physical activity. The behavioral component of the intervention aims to promote walking three to five times per week and is based on the Spanish Projecte Moviment. It will last 12 weeks as this should be sufficient enough to lead to a significant increase in participants' physical activity and cardiorespiratory fitness, and it should also be long enough for physical activity to become an habit. The walking program is based on international guidelines of physical exercise. Participants will be instructed to walk briskly in one continuous bout (45 minutes for 5 days, 225 minutes per week). Intensity, duration, and times per week will be initiated in a stepwise manner to reduce the possibility of injury. During the first week participants will be asked to walk 30 minutes at 9-10 on the Borg Rating of Perceived Exertion Scale (i.e., light intensity). During the second week, participants will be asked to walk 45 minutes with the same intensity. During the remaining weeks, participants will be asked to maintain the duration of 45 minutes and increase the intensity of the activity to a moderate-high effort that corresponds with 12-14 in the Borg Rating of Perceived Exertion Scale. The first day of the psychoeducational intervention participants will be trained to use the Borg Rating of Perceived Exertion Scale and to record this intensity and frequency of activity in a paper daily diary. To ensure adherence to the protocol, every two weeks the project team will contact participants via phone call, text message, or email to check their level of engagement with physical activity and to remind them to record their physical activities in the daily diary.

To anticipate, prevent, and answer medical or personal issues of the participants, the project team will take into account several considerations. First, during an initial screening done via phone, only those participants who are physically fit to start a walking intervention will be allowed to take part in the study (i.e., participants that do not self-report mobility issues and that during the baseline physical fitness assessment do not show any physical concerns/limitations). Second, all the baseline and follow-up assessments will be reviewed by the research team before allocating participants to intervention group to ensure safety during the intervention. Eventual abnormalities identified will be reported and these participants will be directed to corresponding healthcare service. Instructions for the behavioral intervention include healthy advice to prevent injuries. Third, participants can contact the research team for any problems or pain that they may experience. Fourth, to ensure the health and wellbeing of participants throughout the study, every two weeks researchers will also contact participants via text message or email to check whether they are experiencing any physical issues, pain, or if any adverse events occurred while exercising.

Data quality A computerized database will be used to collect and organize all data. Data will be collected without personal identifying information using a code assigned by the researchers. Only the core research team will have access to this information in case of an incident. Data from all participants will be collected/used regardless of whether the participant withdraws from the intervention or not (unless the participant retrospectively asks the study team to destroy their data). All assessments and databases will be double-checked. The study team will follow Data Quality Assessment Checklist and Recommended Procedures that assess a variety of dimensions as validity, reliability, timeliness, precision, and integrity. The study team will analyze whether participants' data is related to expected physical changes. If the study team identifies any issues in the data, they will inform and apply any required statistical procedures to control them.

Statistical analysis To address the first and second study hypotheses, pre-post intervention and follow-up changes in intervention outcomes in the dual-partner intervention group, single-partner intervention group, and control group will be investigated using mixed effects models and/or Structural Equation Modeling. To address the third study hypothesis dyadic mixed effects and/or dyadic structural equation modeling will be used. In all the models, age, sex, education, month when the intervention will be undertaken will be included as covariates. In the models with physical activity as outcome, baseline physical activity will also be included as covariate. To address the third hypothesis, length and quality of the relationship, dominance of the partner, and personality will be considered as additional covariates in the models. Statistical significance level will be set at p < 0.05.

Intention-to-treat analysis will be performed, which means that data of all trial participants in the groups to which they were randomized (i.e., after the collection of baseline data) will be processed, regardless of whether they received or adhered to the allocated intervention. It is assumed that most participants in the first and second groups/arms will receive all intervention sessions. For these analyses, assuming that data is missing at random, missing values will be imputed using multiple imputation by chained equations; 25 imputed datasets will be generated.

Additionally, a per-protocol analysis of the participants who completed the study/intervention without major protocol violation (e.g., who attended at least two of the three psychoeducational sessions and who reported having engaged in physical activity at least 80% of the expected times) will be performed. The per-protocol analysis will be performed as secondary analysis, if there are enough participants in the three intervention groups/arms, who are not lost to follow-up assessments and if there are enough participants in groups one and two who undertook the entirety of the intervention. Quantitative analyses will be conducted using STATA version 19, R, and/or Mplus. Content analysis (111) will be used to analyze data from the open-ended questions and from the interviews conducted at the end of the intervention. These analyses will be conducted using Atlas.ti by two independent researchers.

ELIGIBILITY:
Inclusion criteria are:

* living in the community in Barcelona or nearby areas;
* both partners being aged ≥ 65 years;
* speaking fluent Catalan or Spanish;
* being married, having a partner with whom they co-habit, or having had a partner for at least one year and with whom they meet at least twice a week;
* having access to a smartphone, tablet, laptop, or computer with internet;
* both partners being willing to participate in the study and providing written informed consent.

Although the use of a chronological age cut-off to define older people is inherently arbitrary, this study adopts the threshold of 65 years and older to establish inclusion criteria for participation. This decision reflects the increasing self-relevance of age-stereotypes and self-perceptions of aging in later life, particularly among the oldest age groups. Participants can either possess a device that can be connected to the internet or use the device of a family member, neighbor, or friend. Moreover, participants with low technology literacy can nonetheless take part in the study as during baseline assessment the research team will show them how to complete the online questionnaires. Moreover, the research team will be available via email and phone to answer participants' queries related to completion of the online questionnaires. Both retired and working people are eligible to take part in the study. People of any race can take part in the study. Couples of all sexual orientations are welcome to participate in the study.

Exclusion criteria are:

* having a self-reported or clinically diagnosed neurodegenerative disorder, and/or an Adult Lifestyles and Function Interview Mini Mental State Examination (ALFI-MMSE) score of < 15 out of 22, indicating mild cognitive impairment or dementia. The research team has considerable experience with the administration of the MMSE and will adjust scores for individuals with low cultural background;
* currently having a clinical diagnosis of mental health disorder that significantly impacts on the daily functioning of the individual (i.e., a diagnosis that significantly impacts the participants ability to work, do house chores, and/or engage socially);
* current substance use disorder (alcohol or drug abuse), or a history of substance abuse within the past five years that may interfere with study participation or adherence to the intervention;
* having a physical condition or physical limitations that impair from starting a physical activity intervention consisting in walking between three to five times per week and to do some physical tasks such as stand up from and sit down on a chair and back scratch;
* severe hearing impairment (deafness).

Physical limitations will be self-reported by participants via phone but also further objectively assessed by the researchers at baseline assessment. Individuals with neurodegenerative disorders will be excluded as it could be difficult for them to understand and participate in the psychoeducational sessions, and/or engage in brisk walking. Individuals with current severe mental health disorders and/or with substance abuse will be excluded as these groups are less likely to be compliant with intervention conditions. However, individuals with more common mental health disorders (i.e., depressive disorders and anxiety disorders) that are not severe enough to significantly impact the daily functioning of the individual will be allowed to take part in the study. Individuals with significant physical limitations will be excluded as they could put themselves at risk of falling while engaging in physical activity/walking.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Awareness of Age-Related Change | Baseline, post-intervention (12 weeks after baseline), and three- and six-months follow-ups (post-intervention)
  This 10-item measure assesses self-perceptions of aging. More specifically, it assesses perceived age-related gains and losses. Each of the items of the perceived age-related gains and losses subscales represents one of the five AARC behavioral domains that are health and physical functioning; cognitive functioning; interpersonal relations; social-cognitive and social-emotional functioning; and lifestyle and engagement. Respondents rate how much each item applies to them on a five-point Likert scale (1= not at all; 2= a little bit; 3= moderately; 4= quite a bit; 5= very much). Higher scores indicate higher perceived age-related gains and losses, respectively (range: 5-25).
Felt Age | Baseline, post-intervention (12 weeks after baseline), and three- and six-months follow-ups (post-intervention)
  This measure assesses self-perceptions of aging. Felt age (FA) will be assessed with a single-item question asking participants to write the age (in years) that they feel most of the time. A proportional discrepancy score will be calculated by subtracting the participants' chronological age from their felt age, and by dividing this difference score by participants' chronological age. A positive value indicates an older felt age, whereas a negative value indicates a younger felt age. Typically, in western countries the majority of older individuals feel between 13% and 18% younger than their age, and a younger felt age is used as indicator of more positive self-perceptions of aging.
Subjective Nearness to Death | Baseline, post-intervention (12 weeks after baseline), and three- and six-months follow-ups (post-intervention)
  This measure assesses self-perceptions of aging. Subjective Nearness to Death will be assessed with the one-item question: I have a feeling that my life is approaching its end. Answer options range from 1 (not at all) to 5 (very much).
International Physical Activity Questionnaire | Baseline, post-intervention (12 weeks after baseline), and three- and six-months follow-ups (post-intervention)
  This measure assesses self-reported physical activity. Participants are asked to refer to the past seven days and to report how much time they spent sitting during a day; how many days they walked for at least ten minutes at a time; how many days they did moderate physical activities like gardening, cleaning, and bicycling; and how many days they did vigorous physical activities like heavy lifting, heavier garden or construction work, and aerobics. Separate scores can be obtained for walking, moderate intensity physical activities, and vigorous physical activities as follows: (1) Walking metabolic equivalent of task (MET)-minutes/week = 3.3 * walking minutes * walking days. (2) Moderate MET-minutes/week = 4.0 * moderate-intensity activity minutes * moderate days. (3) Vigorous MET-minutes/week = 8.0 * vigorous-intensity activity minutes * vigorous-intensity days. The International Physical Activity Questionnaire total score derives from the sum of the scores for walking, moderate-inten
Saltin-Grimby Physical Activity Level Scale | Baseline, post-intervention (12 weeks after baseline), and three- and six-months follow-ups (post-intervention)
  This measure assesses self-reported physical activity.The Saltin-Grimby Physical Activity Level Scale consists in a single-item question asking participants to report on average how much they moved during their leisure time. At baseline participants will be asked to answer thinking about the past 12 months whereas at follow-ups they will be asked to think about the past three months. To answer, participants can choose from four categories: 1= physically inactive, 2= some light physical activity, 3= regular physical activity and training, and 4= regular hard physical training for competitive sports.

SECONDARY OUTCOMES:
World Health Organization - Ageism Scale | Baseline, post-intervention (12 weeks after baseline), and three- and six-months follow-ups (post-intervention)
  Experienced ageism will be assessed with 15-items covering self-directed ageism: self-stereotypes (two items), self-prejudice (one item), self-discrimination (two items; interpersonal ageism: interpersonal stereotypes (two items), interpersonal prejudices (two items), interpersonal discrimination (three items) and institutional ageism: institutional discrimination (three items). Answer options for all items are 1= strongly disagree; 2= disagree; 3= neither agree nor disagree; 4= agree; 5= strongly agree. The total score is obtained from the sum of items scores. Higher scores indicate greater ageism.
  Other directed-ageism will be assessed with 23 additional questions developed by the Word Health Organization. Answer options for all items are 1= totally agree; 2= agree; 3= neither agree nor disagree; 4= disagree; 5= strongly disagree. The total score is obtained from the sum of items scores. Higher scores indicate less other-directed ageism.
Subjective Views of Couple's Joint Aging | Baseline, post-intervention (12 weeks after baseline), and three- and six-months follow-ups (post-intervention)
  The 14-item Subjective Views of Couple's Joint Aging (SVoCJA) scale will be used to assess positive and negative subjective views of couple's joint aging. Seven items capture positive subjective views of couple's joint aging and a sample item is the thought that our time together is limited will make us want to love each other more. The remaining seven items capture negative subjective views of couple's joint aging and a sample item is Dealing with health issues will take a heavy toll on our relationship. Each item is answered on a five-point Likert scale: 1= strongly disagree; 2= slightly disagree; 3= neither agree nor disagree; 4= slightly agree; 5= very much agree. Subscales scores are obtained by summing up the scores of their respective items. In the validation sample, Cronbach's alpha coefficients were 0.77 for positive and 0.78 for negative subjective views of couples' joint aging.
Patient Health Questionnaire - 4 | Baseline, post-intervention (12 weeks after baseline), and three- and six-months follow-ups (post-intervention)
  This measure assesses core symptoms of depression and anxiety over the past two weeks. A sample item is Over the last two weeks, how often have you felt little interest or pleasure in doing things? Answer options are on a four-point Likert scale: 1= not at all; 2= several days; 3= more than half the days; 4= nearly every day. The total score is obtained from the sum of items scores. Higher total scores (range: 4-16) indicate more non-specific mood problems. Cronbach's alpha was above 0.80 for both depression and anxiety subscales in the validation sample, indicating good internal reliability.
Body Mass Index | Baseline, post-intervention (12 weeks after baseline), and three- and six-months follow-ups (post-intervention)
  Participants will self-report their height in cm and weight in kg.
Grip Strength | Baseline, post-intervention (12 weeks after baseline), and six-months follow-ups (post-intervention)
  This is an indicator of physical fitness
Senior Fitness Test | Baseline, post-intervention (12 weeks after baseline), and six-months follow-ups (post-intervention)
  It comprises 6 tests. The Chair Stand Test asks participants to repeatedly stand up from and sit down on a chair for 30 sec. The number of stands is recorded. The Biceps Curl Test asks participants to repeatedly lift a 2.27 kg weight for women or an 3.63 kg weight for men for 30 sec. The number of lifts is recorded. The 6-Minute Walk Test asks participants to walk for 6 min on a straight line. The meters walked are recorded. The Chair Sit and Reach Test asks participants to reach forward toward the toes by bending at the hip while being seated. The distance is recorded. The Back Scratch Test asks participants to start from standing position, place one hand behind the head and back over the shoulder and reach as far as possible down the middle of the back and place the other arm behind their back and reach up attempting to touch or overlap the middle fingers of both hands. In the 2.45-m Up-and-Go Test participants stand up from a chair and walk around a cone and to return to the chair.
Trial Making Text A and B | Baseline, post-intervention (12 weeks after baseline), and six-months follow-ups (post-intervention)
  This task assesses cognitive flexibility. Trail Making Test-A requires participants to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper. Task requirements are similar for Trail Making Test-B except the participant must alternate between numbers and letters (e.g., 1, A, 2, B, 3, C, etc.). For both Trail Making Test A and B the total score is the amount of time required to complete the task.
Digit Span Forward and Backward | Baseline, post-intervention (12 weeks after baseline), and six-months follow-ups (post-intervention)
  This task assesses working memory. In the Digit Span Backward participants are asked to repeat digits backward (14 number sequences that range from five to eight digits in length). Each correctly recalled sequence is scored as one point (possible total score range: 0-14). Higher scores indicate greater working memory. In the Digit Span Forward (96) participants are asked to repeat digits forward (14 number sequences ranging from three to nine digits). Each correctly recalled sequence is scored as one point (possible total score range: 0-14). Higher scores indicate greater short-term memory.
PMR Phonological Verbal Fluency Test | Baseline, post-intervention (12 weeks after baseline), and six-months follow-ups (post-intervention)
  This task assesses working memory. In the PMR Phonological Verbal Fluency Test participants are asked to generate within 60 seconds as many words as possible that start with the letters P, M, and R. For each letter the number of correct words is registered, excluding intrusions and perseverations. This task also assesses executive functions in addition to working memory.
Animal Naming Fluency Test | Baseline, post-intervention (12 weeks after baseline), and six-months follow-ups (post-intervention)
  This task assesses working memory. In the Animal Naming Fluency Test participants are asked to generate as many animal names as possible within 60 seconds. This task also assesses executive functions in addition to working memory. The number of correct words is registered, excluding intrusions and perseverations.
Weist circumference | Baseline, three-months follow-up, and 6-months follow-up.
  Waist circumference will be assessed by the researcher during the baseline, post-intervention, and six-month in person follow-up assessments using a flexible measuring tape. The measure will be taken at midpoint between the lower margin of the last palpable rib and the top of the hip bone.
Stroop Color-Word Test | Baseline, three-month follow-up and six-month follow-up. In this test, participants are shown a list of color words, such as "red," "blue," "green", printed in different-colored inks. The ink color may match the word (i.e., congruent condition) or differ
  This task assesses inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Serena Sabatini, PhD in Psychology, Principal Investigator — University of Barcelona
Locations (1):
- Department of Clinical Psychology and Psychobiology at the University of Barcelona., Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared in Open Science Framework once study analyses will have been conducted and the planned publications will have been published.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The study protocol will be available from the start of the project (a detailed protocol will be made available in Open Science Framework). The IPD will be made available at the end of data analyses. We expect tho share IPD by 2028. The analysis plan will be made available at the end of data collection (2027) and the analytic code once data analyses will have been completed (by 2028).
Access Criteria: Everyone will be able to access the anonymised IPD and supporting information via Open Science Framework from 2028.
URL: https://osf.io/wny7f/